CLINICAL TRIAL: NCT05584501
Title: Effectiveness of Comprehensive Ending the Epidemic (ETE) Interventions in the Dental Setting
Brief Title: ETE Interventions in the Dental Setting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAT8854; 1UG3DE031258 (NIH)
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: HIV Infections
Keywords: Health Information Technology; Care Navigation; Acceptability; Feasibility; Dental Setting
MeSH Terms: conditions — HIV Infections | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Each site will experience a care delivery model for 3 months, followed by a 1 month washout period, and then 3 months with the alternative care delivery model.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dental Team (Placebo Comparator): ETE activity implementation with existing Dental Team only (i.e. practitioners, dental assistants, hygienists)
  Interventions: Other: Health Information Supported Ending the HIV Epidemic (ETE) Activities in Dental Setting
- Care Navigator (Active Comparator): ETE activity implementation with additional Care Navigator resource
  Interventions: Other: Care Navigator; Other: Health Information Supported Ending the HIV Epidemic (ETE) Activities in Dental Setting

INTERVENTIONS:
Other: Care Navigator — The Dental Team will have a Care Navigator as an added resource to assist with offering, implementing, and counseling for HIV testing; providing PrEP education and linkage; and providing linkage and re-linkage to HIV care.
  Arms: Care Navigator
Other: Health Information Supported Ending the HIV Epidemic (ETE) Activities in Dental Setting — Dental Teams will receive a Best Practice Alert (BPA) when they have a patient who should be offered HIV testing. Dental Teams will also be notified when they have a patient known to be HIV positive but out of HIV care.

SUMMARY:
The purpose of this study is to use information technology (IT) to support the delivery of HIV prevention and care best practices in the dental care setting to meet the Department of Health and Human Services (DHHS) Ending the HIV Epidemic (ETE) goals.

DETAILED DESCRIPTION:
Routine HIV screening in all health care settings is considered a best practice by the Centers for Disease Control and Prevention (CDC), DHHS Ending the Epidemic Initiative, the New York State Blueprint to End the AIDS Epidemic, and is mandated by law in New York for all individuals over the age of 13 who receive hospital or primary care. Despite this, many patients are not screened for HIV during routine care, including in dental care settings, resulting in missed opportunities for identifying undiagnosed HIV infections, providing education for and linkage to PrEP, and linking and re-engaging HIV-positive patients into HIV care. The investigators will use information technology in the following two ways to support the delivery of HIV prevention and care best practices in the dental care setting to meet the DHHS Ending the HIV Epidemic (ETE) goals. First, Dental Teams will receive a Best Practice (BPA) alert whenever they have a patient who should be offered HIV testing. This BPA is linked to an order set to simplify ordering HIV tests and reporting results. Second, Dental teams will be contacted whenever they have a patient who is known to have HIV and is out of HIV care. A critical knowledge gap for implementing these ETE activities in the dental setting is whether comprehensive ETE efforts could be integrated into existing dental teams consisting of practitioners, dental assistants and hygienists or require augmentation by a dedicated care navigator. Therefore the investigators will pilot the Dental Team and Care Navigator models at two different dental sites (NYP-Columbia and NYP-Weill Cornell) using a cross-over design to evaluate acceptability and feasibility of providing HIV prevention and treatment services supported by these health IT strategies in the dental setting under these two care delivery models. If the strategies are found to be acceptable and feasible for both dental care patients and providers, then the study will expand to 4 sites and examine the effectiveness of these strategies for delivering HIV prevention and care best practices in the dental setting.

ELIGIBILITY:
Inclusion Criteria:

Dental Team/Patient Navigator:

To be eligible, members of the Dental Team or Patient Navigator need to have direct contact with patients at a participating dental clinic site during the months of the pilot study.

Patient:

To be eligible, patients must:

* Be 18 years or older
* Have at least one visit during the months of the pilot study at a participating dental clinic

Exclusion Criteria:

* Not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Acceptability among Patients | Within 2 weeks after the patient's dental visit
  Acceptability of the intervention under the two arms will be assessed using the validated Acceptability of Intervention Measure (AIM). AIM is a 4-item scale where respondents rate each item using a 5-point ordinal scale that ranges from "completely disagree=1" to "completely agree=5". The AIM is scored by averaging responses across the 4 items. A higher average score indicates greater acceptability, which is a better outcome.
Acceptability among Providers | Within 2 weeks after the patient's dental visit
  Acceptability of the intervention under the two arms will be assessed using the validated Acceptability of Intervention Measure (AIM). AIM is a 4-item scale where respondents rate each item using a 5-point ordinal scale that ranges from "completely disagree=1" to "completely agree=5". The AIM is scored by averaging responses across the 4 items. A higher average score indicates greater acceptability, which is a better outcome.
Feasibility among Providers | Within 9 months from baseline
  Feasibility of the intervention under the two arms will be assessed using the validated Feasibility of Intervention Measure (FIM). FIM is a 4-item scale where respondents rate each item using a 5-point ordinal scale that ranges from "completely disagree=1" to "completely agree=5". The FIM is scored by averaging responses across the 4 items. A higher average score indicates greater feasibility, which is a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Yin, MD, MS, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Irving Medical Center / NewYork-Presbyterian Hospital, New York, New York
  - Weill Cornell Medical Center / NewYork-Presbyterian Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data may be shared with other researchers within Columbia University at the discretion of the Principal Investigator, and only when the Institutional Review Board (IRB) approval has been granted to allow for the sharing of such data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data and supporting information will be made available no later than the acceptance for publication of the main findings from the final dataset.
Access Criteria: At the discretion of the Principal Investigator, and only when the Institutional Review Board (IRB) approval has been granted to allow for the sharing of such data.